CLINICAL TRIAL: NCT03130569
Title: Personalized Genomic Testing for Skin Cancer - Maximizing Utility and Reach
Brief Title: Skin Health Online for Melanoma: Better Risk Assessment
Acronym: SOMBRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, Marianne Berwick, Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-050
Record Dates: First submitted 2017-04-19; First posted 2017-04-26 (Actual); Results first posted 2024-11-18 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Melanoma (Skin)
Keywords: Risk Assessment; Personal Genomic Testing; Skin Cancer; Primary Care
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Will simply complete surveys at baseline and at the three-month follow-up.
- Web-based Module Group (Experimental): Participants will complete surveys at baseline. Participants in this arm will be provided with information to access and complete a web-based educational module (AKA the intervention), at the end of which will be given the opportunity to request and complete genetic testing for skin cancer. Participants who elect to complete the genetic testing will receive their genetic testing results along with a two-week follow-up call. All participants will also complete the survey at the three month follow-up.
  Interventions: Behavioral: Web-based Module Group

INTERVENTIONS:
Behavioral: Web-based Module Group
  Arms: Web-based Module Group

SUMMARY:
This study will have two phases, with an added usability test after Phase I and before Phase 2. Phase 1: Cognitive Interviews of materials in Spanish. Phase 2: Personalized Genomic Testing for Skin Cancer (PGT-SC). The overarching goal of this study is to learn more about how to maximize the availability, comprehension and appropriate uptake of personalized genomics among different populations in New Mexico. Primary Care patients will be recruited in their primary health clinic to complete surveys about their understanding and beliefs of skin cancer and behaviors that might help prevent skin cancer. 6 out of every 7 patients will then be asked to go to a website to learn more about skin cancer risk. Once participants have completed the education modules on this site, participants will be given the option to request and complete a skin cancer genetic testing kit. All participants will be contacted again after three months to complete a follow-up set of surveys about skin cancer.

DETAILED DESCRIPTION:
This study will have two phases, with an added usability test after Phase I and before Phase 2. Phase 1: Cognitive Interviews in Spanish. Phase 2: Personalized Genomic Testing for Skin Cancer (PGT-SC).

The overarching goal of this study is to learn more about how to maximize the availability, comprehension and appropriate uptake of personalized genomics among different populations in New Mexico. The study has been funded as an R01 by NCI for three years.

Aim I: To examine the personal utility (that is, how does personal genomic testing help the individual) of Personal Genomic Testing for Skin Cancer (PGT-SC) in terms of short-term (three months after testing) sun protection, skin screening (i.e., behaviors), communication, melanoma threat and control beliefs (i.e., putative mediators of behavior change). Guided by Protection Motivation Theory, the investigators hypothesize that behaviors and putative mediators will be higher in those who test, compared to those who decline testing or wait-list controls.

Aim Ia. An important challenge of personal genomics involves the potential for those who receive "negative" genetic feedback to increase risky behaviors. To examine this potential unintended consequence of testing, the investigators will conduct a subgroup analysis among those who receive average risk PGT-SC findings, examining sun protection at three months as the outcome. Predictors will include baseline skin cancer threat and control beliefs, skin cancer risk factors, and demographics. These findings will be used in future studies to develop messages for groups that receive average risk feedback, which accounts for large segments of those tested for moderate risk susceptibility factors across many diseases.

Aim II: To examine differential reach of PGT-SC across Hispanics and Non-Hispanics, and potential explanations for any differential reach. Reach is defined as the extent to which genomic testing is spread throughout the population. Reach will be measured in individuals as the consideration of the pros and cons of testing and registration of test decision. Additional assessments of reach include baseline survey completion and decision to pursue PGT-SC testing. The investigators hypothesize that those who are self-identified Hispanic will show reduced reach, but that differences in health literacy, health system distrust, and Hispanic sociocultural factors including cancer fatalism, family health orientation, and skin cancer misperceptions will explain differences in reach between Hispanics and Non-Hispanics, and provide guidance for future PGT-SC modifications for Hispanics.

Aim III: Among those who undergo testing, to examine (two weeks after PGT-SC test result receipt) test comprehension, recall, satisfaction, and cancer-related distress, and whether these outcomes differ by ethnicity (Hispanic versus Non-Hispanic) or health literacy, distrust, sociocultural, or demographic factors. The investigators hypothesize, based on prior work delivering this intervention in primary care, the results will reflect high test comprehension, accurate feedback interpretation, and low test distress in those who get tested.

Background. Personalized genomics currently has extremely limited reach. First, most gene discovery has not engaged diverse research cohorts. Second, the few translational research efforts that address "real world" genomic challenges and opportunities have engaged those with higher socioeconomic status and health literacy. Third, ethnic and racial minorities are less likely to participate in basic genomics research, and are also less likely to utilize available genomic technologies, even when they are offered. Ideally, the investigators should all have fair access to the knowledge gained from sequencing the human genome, but if these trends continue, the investigators will know little about how to maximize availability, comprehension, and appropriate uptake of personalized genomics across large subpopulations that stand to benefit from it.

To begin to address this, The Multiplex Study led by the National Human Genome Research Institute (NHGRI) used population-based recruitment strategies in Detroit, Michigan to evaluate an Internet-provided offer of genomic testing for common diseases, including melanoma, the most serious form of skin cancer. Study findings indicate that this approach is feasible - resulting in high test comprehension, accurate feedback interpretation, and low test distress in those who sought testing. Yet this study did not include Hispanics nor assess behavioral outcomes.

Personalized genomic testing for skin cancer (PGT-SC) is an ideal context to extend Multiplex to a new population, and new outcomes. Skin cancers are preventable, curable, very common in the general population, and disproportionately increasing in Hispanics. The NHGRI Multiplex Study offered testing for melanoma risk via the melanocortin 1 receptor gene (MC1R) because MC1R is common in the general population (50% >1 high risk variant), interacts with sun exposure, and confers risk (2-3 fold; consistent with most moderate risk variants), even in those with darker skin types. MC1R feedback is a promising vehicle to raise risk awareness and protective behavior in the general population, including Hispanics who are largely unaware of their melanoma risks. The investigators will conduct a randomized controlled trial examining internet presentation of the risks and benefits of PGT-SC (shown to be feasible in Multiplex) versus wait-list controls who are not offered testing, comparing personal utility and reach in a general population, English or Spanish-speaking cohort in Albuquerque, New Mexico, where there is year-round sun exposure.

Phase 1 data is not reported in the Results section because the goal of Phase 1 was to finalize the Spanish translation of the intervention/data collection instruments.

ELIGIBILITY:
Inclusion Criteria:

* Registered at a University of New Mexico primary care clinic for ≥6 months
* Assigned to a primary care provider
* Fluent in either English or Spanish

Exclusion Criteria:

* Unable to consent
* <18 years old
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Berwick, PhD, Principal Investigator — University of New Mexico; Jennifer Hay, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloss CS, Ornowski L, Silver E, Cargill M, Vanier V, Schork NJ, Topol EJ. Consumer perceptions of direct-to-consumer personalized genomic risk assessments. Genet Med. 2010 Sep;12(9):556-66. doi: 10.1097/GIM.0b013e3181eb51c6. PMID 20717041
- [Background] Demenais F, Mohamdi H, Chaudru V, Goldstein AM, Newton Bishop JA, Bishop DT, Kanetsky PA, Hayward NK, Gillanders E, Elder DE, Avril MF, Azizi E, van Belle P, Bergman W, Bianchi-Scarra G, Bressac-de Paillerets B, Calista D, Carrera C, Hansson J, Harland M, Hogg D, Hoiom V, Holland EA, Ingvar C, Landi MT, Lang JM, Mackie RM, Mann GJ, Ming ME, Njauw CJ, Olsson H, Palmer J, Pastorino L, Puig S, Randerson-Moor J, Stark M, Tsao H, Tucker MA, van der Velden P, Yang XR, Gruis N; Melanoma Genetics Consortium. Association of MC1R variants and host phenotypes with melanoma risk in CDKN2A mutation carriers: a GenoMEL study. J Natl Cancer Inst. 2010 Oct 20;102(20):1568-83. doi: 10.1093/jnci/djq363. Epub 2010 Sep 28. PMID 20876876
- [Background] Friedman LC, Bruce S, Weinberg AD, Cooper HP, Yen AH, Hill M. Early detection of skin cancer: racial/ethnic differences in behaviors and attitudes. J Cancer Educ. 1994 Summer;9(2):105-10. doi: 10.1080/08858199409528281. PMID 7917894
- [Background] Green ED, Guyer MS; National Human Genome Research Institute. Charting a course for genomic medicine from base pairs to bedside. Nature. 2011 Feb 10;470(7333):204-13. doi: 10.1038/nature09764. PMID 21307933
- [Background] Hay J, Ostroff J, Martin A, Serle N, Soma S, Mujumdar U, Berwick M. Skin cancer risk discussions in melanoma-affected families. J Cancer Educ. 2005 Winter;20(4):240-6. doi: 10.1207/s15430154jce2004_13. PMID 16497137
- [Background] Hay J, Shuk E, Brady MS, Berwick M, Ostroff J, Halpern A. Family communication after melanoma diagnosis. Arch Dermatol. 2008 Apr;144(4):553-4. doi: 10.1001/archderm.144.4.553. No abstract available. PMID 18427057
- [Background] Hay J, Shuk E, Zapolska J, et al. Family communication patterns after melanoma diagnosis. Journal of Family Communication. 2009;9(4):209-232.
- [Background] Hay J, Coups EJ, Ford J, DiBonaventura M. Exposure to mass media health information, skin cancer beliefs, and sun protection behaviors in a United States probability sample. J Am Acad Dermatol. 2009 Nov;61(5):783-92. doi: 10.1016/j.jaad.2009.04.023. Epub 2009 Jul 10. PMID 19596487
- [Background] Hay JL, Baguer C, Li Y, Orlow I, Berwick M. Interpretation of melanoma risk feedback in first-degree relatives of melanoma patients. J Cancer Epidemiol. 2012;2012:374842. doi: 10.1155/2012/374842. Epub 2012 Jul 25. PMID 22888347
- [Background] Hay J, Kaphingst KA, Baser R, Li Y, Hensley-Alford S, McBride CM. Skin cancer concerns and genetic risk information-seeking in primary care. Public Health Genomics. 2012;15(2):57-72. doi: 10.1159/000330403. Epub 2011 Sep 13. PMID 21921576
- [Background] Hindorff LA, Sethupathy P, Junkins HA, Ramos EM, Mehta JP, Collins FS, Manolio TA. Potential etiologic and functional implications of genome-wide association loci for human diseases and traits. Proc Natl Acad Sci U S A. 2009 Jun 9;106(23):9362-7. doi: 10.1073/pnas.0903103106. Epub 2009 May 27. PMID 19474294
- [Background] Hu S, Parmet Y, Allen G, Parker DF, Ma F, Rouhani P, Kirsner RS. Disparity in melanoma: a trend analysis of melanoma incidence and stage at diagnosis among whites, Hispanics, and blacks in Florida. Arch Dermatol. 2009 Dec;145(12):1369-74. doi: 10.1001/archdermatol.2009.302. PMID 20026844
- [Background] James RD, Yu JH, Henrikson NB, Bowen DJ, Fullerton SM; Health Disparities Working Group. Strategies and stakeholders: minority recruitment in cancer genetics research. Community Genet. 2008;11(4):241-9. doi: 10.1159/000116878. Epub 2008 Apr 14. PMID 18417972
- [Background] Kaphingst KA, McBride CM, Wade C, Alford SH, Reid R, Larson E, Baxevanis AD, Brody LC. Patients' understanding of and responses to multiplex genetic susceptibility test results. Genet Med. 2012 Jul;14(7):681-7. doi: 10.1038/gim.2012.22. PMID 22481132
- [Background] Khoury MJ, Clauser SB, Freedman AN, Gillanders EM, Glasgow RE, Klein WM, Schully SD. Population sciences, translational research, and the opportunities and challenges for genomics to reduce the burden of cancer in the 21st century. Cancer Epidemiol Biomarkers Prev. 2011 Oct;20(10):2105-14. doi: 10.1158/1055-9965.EPI-11-0481. Epub 2011 Jul 27. PMID 21795499
- [Background] Lazovich D, Choi K, Vogel RI. Time to get serious about skin cancer prevention. Cancer Epidemiol Biomarkers Prev. 2012 Nov;21(11):1893-901. doi: 10.1158/1055-9965.EPI-12-0327. Epub 2012 Sep 7. PMID 22962407
- [Background] Mujumdar UJ, Hay JL, Monroe-Hinds YC, Hummer AJ, Begg CB, Wilcox HB, Oliveria SA, Berwick M. Sun protection and skin self-examination in melanoma survivors. Psychooncology. 2009 Oct;18(10):1106-15. doi: 10.1002/pon.1510. PMID 19142859
- [Background] Pagan JA, Su D, Li L, Armstrong K, Asch DA. Racial and ethnic disparities in awareness of genetic testing for cancer risk. Am J Prev Med. 2009 Dec;37(6):524-30. doi: 10.1016/j.amepre.2009.07.021. PMID 19944919
- [Background] Pipitone M, Robinson JK, Camara C, Chittineni B, Fisher SG. Skin cancer awareness in suburban employees: a Hispanic perspective. J Am Acad Dermatol. 2002 Jul;47(1):118-23. doi: 10.1067/mjd.2002.120450. PMID 12077590
- [Background] Raimondi S, Sera F, Gandini S, Iodice S, Caini S, Maisonneuve P, Fargnoli MC. MC1R variants, melanoma and red hair color phenotype: a meta-analysis. Int J Cancer. 2008 Jun 15;122(12):2753-60. doi: 10.1002/ijc.23396. PMID 18366057
- [Background] Robinson JK, Joshi KM, Ortiz S, Kundu RV. Melanoma knowledge, perception, and awareness in ethnic minorities in Chicago: recommendations regarding education. Psychooncology. 2011 Mar;20(3):313-20. doi: 10.1002/pon.1736. PMID 20878831
- [Background] Rouhani P, Pinheiro PS, Sherman R, Arheart K, Fleming LE, Mackinnon J, Kirsner RS. Increasing rates of melanoma among nonwhites in Florida compared with the United States. Arch Dermatol. 2010 Jul;146(7):741-6. doi: 10.1001/archdermatol.2010.133. PMID 20644034
- [Background] Suther S, Kiros GE. Barriers to the use of genetic testing: a study of racial and ethnic disparities. Genet Med. 2009 Sep;11(9):655-62. doi: 10.1097/GIM.0b013e3181ab22aa. PMID 19752639
- [Background] Torres S, Ramos M, Leverence R, Bowen D, Berwick M, Hay J. Skin Cancer Risk Reduction Behaviors, Cancer Communication, and Skin Cancer Beliefs in Hispanics in a Southwestern Primary Care Practice. Californian Journal of Health Promotion. See Appendix III for the In Press Manuscript.
- [Background] Udayakumar D, Tsao H. Moderate- to low-risk variant alleles of cutaneous malignancies and nevi: lessons from genome-wide association studies. Genome Med. 2009 Oct 27;1(10):95. doi: 10.1186/gm95. PMID 19863770
- [Background] Wade CH, McBride CM, Kardia SL, Brody LC. Considerations for designing a prototype genetic test for use in translational research. Public Health Genomics. 2010;13(3):155-65. doi: 10.1159/000236061. Epub 2009 Sep 3. PMID 19729884
- [Derived] Hay JL, Zielaskowski K, Meyer White K, Kaphingst K, Robers E, Guest D, Sussman A, Talamantes Y, Schwartz M, Rodriguez VM, Li Y, Schofield E, Bigney J, Hunley K, Buller D, Berwick M. Interest and Uptake of MC1R Testing for Melanoma Risk in a Diverse Primary Care Population: A Randomized Clinical Trial. JAMA Dermatol. 2018 Jun 1;154(6):684-693. doi: 10.1001/jamadermatol.2018.0592. PMID 29801061

RESULTS

PARTICIPANT FLOW:
Groups:
- Web-based Module Group: Participants will complete surveys at baseline. Participants in this arm will be provided with information to access and complete a web-based educational module (AKA the intervention), at the end of which will be given the opportunity to request and complete genetic testing for skin cancer. Participants who elect to complete the genetic testing will receive their genetic testing results along with a two-week follow-up call. All participants will also complete the survey at the three month follow-up.
  Web-based Module Group
Period: Overall Study
Arm/Group | Control Group | Web-based Module Group
Started | 101 | 499
Completed | 82 | 401
Not Completed | 19 | 98

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Web-based Module Group | Total
Number analyzed (Participants) | 101 | 499 | 600
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 377 | 454
  >=65 years | 23 | 115 | 138
  Unknown or Not Reported | 1 | 7 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 396 | 473
  Male | 24 | 103 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 242 | 286
  Not Hispanic or Latino | 57 | 255 | 312
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian / Alaska Native | 2 | 13 | 15
  Asian | 1 | 11 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 2 | 13 | 15
  White | 67 | 356 | 423
  More than 1 race | 8 | 13 | 21
  Other race | 20 | 91 | 111
  Unknown race | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 101 | 499 | 600

OUTCOME MEASURES:

1. Primary Outcome: Reach of Personalized Genomic Testing for Melanoma.
Description: Reach is defined as registration of a personalized genomic testing for melanoma (PGT-M) test decision, either for or against testing (dichotomous outcome; test decision or no test decision). Additional assessments of reach include baseline survey completion and decision to pursue PGT-M testing.
Time Frame: Three months from enrollment for each participant. Enrollment occurs on a rolling basis, to be completed August 2017.
Population: Data for this outcome was not collected for the control group.
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Group that received no intervention
- Web-Based Module Group: Group that completed the web-based modules and were offered the opportunity to test.
Arm/Group | Control Group | Web-Based Module Group
Number analyzed (Participants) | 0 | 499
Participants
  Registered a Test Decision For Testing | 0 | 204
  Registered a Test Decision Against Testing | 0 | 295

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Control Group | Web-based Module Group
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/499
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/499
Other Adverse Events (participants affected / at risk) | 0/101 | 0/499

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT03130569/Prot_SAP_000.pdf